CLINICAL TRIAL: NCT02337738
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 2/3 Study to Evaluate the Efficacy and Safety of TVP-1012 at 0.5 mg or 1 mg in Levodopa Treated Parkinson's Disease Patients With Wearing Off
Brief Title: A Phase 2/3 Study of TVP-1012 at 0.5 mg or 1 mg in Levodopa Treated Parkinson's Disease Participants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVP-1012/CCT-002; U1111-1165-1364 (Registry Identifier: WHO); JapicCTI-152759 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TVP-1012 1mg (Experimental): TVP-1012 1 mg once daily orally, before or after breakfast, concomitantly with levodopa tablet for 26 weeks as treatment period after 2 weeks of run-in period.
  Interventions: Drug: TVP-1012 1mg
- TVP-1012 0.5mg (Experimental): TVP-1012 0.5 mg once daily orally, before or after breakfast, concomitantly with levodopa tablet for 26 weeks as treatment period after 2 weeks of run-in period.
  Interventions: Drug: TVP-1012 0.5mg
- Placebo (Placebo Comparator): One placebo tablet once daily orally, before or after breakfast, concomitantly with levodopa tablet for 26 weeks as treatment period after 2 weeks of run-in period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TVP-1012 1mg — TVP-1012 1mg Tablets
  Arms: TVP-1012 1mg
Drug: TVP-1012 0.5mg — TVP-1012 0.5mg Tablets
  Arms: TVP-1012 0.5mg
Drug: Placebo — Placebo Tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TVP-1012 (0.5 mg or 1 mg/day) as an add-on to levodopa in Japanese participants with Parkinson's disease with wearing-off phenomenon.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, phase 2/3 study to evaluate the efficacy and safety of TVP-1012 as an add-on to levodopa in Japanese participants with Parkinson's disease with wearing-off phenomenon.

The study period consisted of a 28-week trial period. The participants who fulfilled the inclusion criteria and did not meeting any of the exclusion criteria were enrolled, and randomized in a 1:1:1 ratio to the 0.5 mg of TVP-1012, the 1 mg of TVP-1012, or the placebo group. In each treatment group, participants received 0.5 mg of TVP-1012, 1 mg of TVP-1012, or placebo once daily in a double-blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
* The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* The participant has a diagnosis of Parkinson's disease according to the diagnostic criteria of the UK Parkinson's Disease Society Brain Bank.
* The participant has Modified Hoehn & Yahr stage 2 to 4 (in the "Off" state) at the start of the run-in period.
* The participant has wearing off phenomenon and has been continuously receiving a levodopa combination drug for >= 6 months prior to the start of the run-in period.
* The participant has been receiving a levodopa combination drug with a stable dose regimen (dosing frequency, at least 3 times a day) since the start of the run-in period.
* For participants receiving eantacapone concomitantly,the participant has been receiving entacapone with a stable dose regimen from the start of the run-in period.
* For participants receiving a dopamine agonist, anticholinergic drug, amantadine, droxidopa, istradefylline, or zonisamide concomitantly, the participant has been receiving those drugs with a stable dose regimen since 14 days prior to the start of the run-in period.
* The participant is an outpatient of either sex aged >= 30 and < 80 years at the time of consent.
* A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent to 1 month after the last dose of the investigational drug.
* The participant has completed patient diary for at least 4 of the 7 days preceding the study visit at the end of the run-in period.
* The participant has mean daily off-time of >= 2.5 hours at the end of the run-in period

Exclusion Criteria:

* The participant has received any investigational medication within 90 days prior to the start of the run-in period.
* The participant has received TVP-1012 in the past.
* The participant is a study site employee, an immediate family member, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
* Participant has donated 400 mL or more of his or her blood volume within 90 days prior to the start of the run-in period.
* The participant has unstable systemic disease.
* The participant has severe dyskinesia.
* The participant has Mini-Mental State Examination (MMSE) score of <= 24 at the start of the run-in period.
* The participant has known or a history of schizophrenia, major or severe depression, or any other clinically significant psychiatric disease
* The participant has major depression or severe depression, or any other clinically significant psychiatric disease.
* The participant has a history of hypersensitivity or allergies to TVP-1012 (including any associated excipients) or selegiline.
* The participant has a history of clinically significant hypertension or other reactions associated with ingestion of tyramine-rich food (e.g., cheese, lever, herring, yeast, horsebean, banana, beer or wine).
* The participant has a history or concurrent of drug abuse or alcohol dependence.
* The participant has received neurosurgical intervention for Parkinson's disease (e.g., pallidotomy, thalamotomy, deep brain stimulation).
* The participant has received transcranial magnetic stimulation within 6 months prior to the start of the run-in period.
* The participant has received selegiline, pethidine, tramadol, reserpine or methyldopa within 90 days prior to the start of the run-in period.
* The participant has received single agent of levodopa, any psychoneurotic agent or antiemetic medication of dopamine antagonist within 14 days prior to the start of the run-in period. However, the participant has been receiving quetiapine or domperidone with a stable dose regimen for >= 14 days prior to the start of the run-in period may be included in the study.
* The participant is required to take any of the prohibited concomitant medications or treatments.
* If female, the participant is pregnant or lactating or intending to become pregnant during, or within 1 month after the last administration of study medication in this study; or intending to donate ova during such time period.
* The participant has clinically significant neurologic, cardiovascular, pulmonary, hepatic (including mild cirrhosis), renal, metabolic, gastrointestinal, urological, endocrine, or hematological disease.
* The participant has clinically significant or unstable brain or cardiovascular disease, such as:

  * clinically significant arrhythmia or cardiac valvulopathy,
  * heart failure of NYHA Class II or higher,
  * concurrent or a history of ischemic cardiac disease within 6 months prior to the start of the run-in period,
  * concurrent or a history of clinically significant cerebrovascular disease within 6 months prior to the stat of the run-in period,
  * severe hypertension (systolic blood pressure of 180 mmHg or higher, or diastolic blood pressure of 110 mmHg or higher),
  * clinically significant orthostatic hypotension (including those with diastolic pressure decrease of 30 mmHg or more following postural change from supine/sitting position to standing position), or
  * a history of syncope due to hypotension within 2 years prior to the stat of the run-in period.
* The participant is required surgery or hospitalization for surgery during the study period.
* Participant has a history of cancer within 5 years prior to the start of the run-in period, except cervix carcinoma in situ which has completely cured.
* The participant has acquired immunodeficiency syndrome (AIDS) [including human immunodeficiency virus (HIV) carrier], or hepatitis [including viral hepatitis carrier such as hepatitis B surface (HBs) antigen or hepatitis C antibody (HCV) positive]. However, the participant who has a negative result for HCV antigen or HCV-RNA can be included in the study.
* The participant has laboratory data meeting any of the following at the start of the run-in period:

  * Creatinine >= 2 x upper limit of normal (ULN)
  * Total bilirubin >= 2 x ULN
  * ALT or AST >= 1.5 x ULN
  * ALP >= 3 x ULN
* The participant has received any of the prohibited concomitant medications or treatments during the run-in period.
* The participant who, in the opinion of the investigator or sub-investigator, is unsuitable for any other reason.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2016-09-17 (Actual); Study Completion 2016-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (57):
- Japan (57):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Touon, Ehime
  - Kitakyushu, Fukuoka
  - Onoshiro, Fukuoka
  - Aizu-Wakamatsu, Fukushima
  - Fujioka, Gunma
  - Asahikawa, Hokkaido
  - Iwamizawa, Hokkaido
  - Sapporo, Hokkaido
  - Akashi, Hyōgo
  - Kobe, Hyōgo
  - Tsukuba, Ibaragi
  - Morioka, Iwate
  - Takamatsu, Kagawa-ken
  - Fujisawa, Kanagawa
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Nankoku, Kochi
  - Gōshi, Kumamoto
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Higashisonogi-gun, Nagasaki
  - Jōetsu, Niigata
  - Yufu, Oita Prefecture
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Toyonaka, Osaka
  - Irima-gun, Saitama
  - Fuji, Shizuoka
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Shimono, Tochigi
  - Yoshinogawa, Tokushima
  - Bunkyo-ku, Tokyo
  - Fuchū, Tokyo
  - Kodaira, Tokyo
  - Nerima-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Akita
  - Aomori
  - Chiba
  - Fukuoka
  - Fukushima
  - Hiroshima
  - Kyoto
  - Miyazaki
  - Niigata
  - Okayama
  - Osaka
  - Tokushima
  - Toyama
  - Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hattori N, Takeda A, Hanya Y, Kitagawa T, Arai M, Furusawa Y, Mochizuki H, Nagai M, Takahashi R. Effects of rasagiline on Parkinson's Disease Questionnaire (PDQ-39) emotional well-being domain in patients with Parkinson's disease: A post-hoc analysis of clinical trials in Japan. PLoS One. 2022 Jan 25;17(1):e0262796. doi: 10.1371/journal.pone.0262796. eCollection 2022. PMID 35077474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 68 investigative sites in Japan, from 27-Jan-2015 to 15-Sep-2016.
Pre-assignment Details: Participants with diagnosis of Parkinson's disease with wearing-off phenomenon who were enrolled in run- in period (Week -2 to 0). After that, the participants who fulfilled the inclusion criteria and did not meet any of the exclusion criteria at Week -2 and Week 0 were randomized in 1:1:1 to TVP-1012 0.5 mg, TVP-1012 1 mg, or placebo at Week 0.
Groups:
- Placebo: For 2 weeks during the run-in period, followed by 26 weeks during the treatment period, one placebo tablet once daily orally, either before or after breakfast, concomitantly with levodopa tablet
- TVP-1012 0.5 mg: For 2 weeks during the run-in period, followed by 26 weeks during the treatment period, TVP-1012 0.5 mg once daily orally, either before or after breakfast, concomitantly with levodopa tablet
- TVP-1012 1 mg: For 2 weeks during the run-in period, followed by 26 weeks during the treatment period, TVP-1012 1 mg once daily orally, either before or after breakfast, concomitantly with levodopa tablet
Period: Overall Study
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Started | 141 | 134 | 129
Completed | 119 | 104 | 103
Not Completed | 22 | 30 | 26
Not completed — Major Protocol Deviation (Pre-Treatment) | 0 | 1 | 0
Not completed — Pretreatment Event/Adverse Event | 9 | 18 | 21
Not completed — Major Protocol Deviation (in-Treatment) | 0 | 1 | 0
Not completed — Voluntary Withdrawal | 10 | 5 | 2
Not completed — Lack of Efficacy | 2 | 4 | 0
Not completed — Investigator's Judgment | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Randomized set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg | Total
Number analyzed (Participants) | 141 | 134 | 129 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.62) | 66.1 (8.74) | 65.8 (8.48) | 66.1 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 76 | 83 | 247
  Male | 53 | 58 | 46 | 157
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan: Japan | 141 | 134 | 129 | 404
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 156.7 (9.61) | 157.1 (10.49) | 156.6 (8.78) | 156.8 (9.64)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 54.30 (12.723) | 56.54 (12.545) | 54.23 (11.762) | 55.02 (12.377)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 21.99 (3.917) | 22.87 (4.049) | 21.98 (3.584) | 22.28 (3.871)
Smoking Classification [Count of Participants; unit: Participants]
  Current Smoker | 5 | 12 | 10 | 27
  Ex-Smoker | 41 | 43 | 34 | 118
  Never Smoked | 95 | 79 | 85 | 259
Timing of Study Drug Dose [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 141 | 133 | 129 | 403
    Before Breakfast | 68 | 61 | 67 | 196
    After Breakfast | 73 | 72 | 62 | 207
Duration of Parkinson's Disease [Mean (Standard Deviation); unit: years] | 8.90 (4.465) | 8.53 (4.774) | 9.49 (4.992) | 8.96 (4.745)
Duration of Levodopa Use [Mean (Standard Deviation); unit: years] | 6.49 (4.402) | 5.94 (3.984) | 7.17 (4.800) | 6.53 (4.420)
Levodopa Total Daily Dose [Mean (Standard Deviation); unit: mg per day] | 399.3 (141.03) | 407.8 (134.15) | 420.7 (166.42) | 409.0 (147.48)
Levodopa Frequency per Day [Mean (Standard Deviation); unit: times per day] | 3.8 (1.07) | 3.9 (1.32) | 4.1 (1.38) | 3.9 (1.26)
Concomitant Use of COMT Inhibitor [Count of Participants; unit: Participants] — COMT; catechol-O-methyltransferase
  Participants
    Had COMT Inhibitor | 54 | 59 | 54 | 167
    Had no COMT Inhibitor | 87 | 75 | 75 | 237
Concomitant Use of Dopamine Agonist [Count of Participants; unit: Participants]
  Had Dopamine Agonist | 122 | 106 | 114 | 342
  Had no Dopamine Agonist | 19 | 28 | 15 | 62
Concomitant Use of Amantadine [Count of Participants; unit: Participants]
  Had Amantadine | 23 | 26 | 33 | 82
  Had no Amantadine | 118 | 108 | 96 | 322
Concomitant Use of Anticholinergics [Count of Participants; unit: Participants]
  Had Anticholinergics | 12 | 13 | 13 | 38
  Had no Anticholinergics | 129 | 121 | 116 | 366
Concomitant Use of Droxidopa [Count of Participants; unit: Participants]
  Had Droxidopa | 8 | 11 | 11 | 30
  Had no Droxidopa | 133 | 123 | 118 | 374
Concomitant Use of Istradefylline [Count of Participants; unit: Participants]
  Had Istradefylline | 33 (2.869) | 24 (2.749) | 35 (2.990) | 92
  Had no Istradefylline | 108 | 110 | 94 | 312
Concomitant Use of Zonisamide [Count of Participants; unit: Participants]
  Had Zonisamide | 45 (0.608) | 51 (0.542) | 52 (0.566) | 148
  Had no Zonisamide | 96 | 83 | 77 | 256
Duration of Wearing Off Phenomenon [Mean (Standard Deviation); unit: years] | 2.94 (2.869) | 2.89 (2.749) | 3.27 (2.990) | 3.03 (2.867)
Modified Hoehn & Yahr Stage (ON State) [Mean (Standard Deviation); unit: Units on a scale] — Modified Hoehn & Yahr Stage represented severity for symptoms of Parkinson's disease progress. The Stage of Modified Hoehn & Yahr were assigned from Stage 0 (Asymptomatic) to Stage 5 (Wheelchair bound or bedridden unless aided (unable to walk even if aided)). ON-state refers to periods of the day when levodopa is working well.
  Units on a scale | 2.44 (0.608) | 2.45 (0.542) | 2.51 (0.566) | 2.46 (0.573)
Modified Hoehn & Yahr Stage (OFF State) [Mean (Standard Deviation); unit: Units on a scale] — Modified Hoehn & Yahr Stage represented severity for symptoms of Parkinson's disease progress. The Stage of Modified Hoehn & Yahr were assigned from Stage 0 (Asymptomatic) to Stage 5 (Wheelchair bound or bedridden unless aided (unable to walk even if aided)). OFF-state refers to periods of the day when levodopa is not working well.
  Units on a scale | 3.22 (0.708) | 3.25 (0.674) | 3.30 (0.651) | 3.26 (0.678)
Mean Daily OFF-time [Mean (Standard Deviation); unit: hours per day] — Off-time refers to times when levodopa is not working well, causing worsening symptoms.
  hours per day | 6.05 (2.278) | 6.33 (2.562) | 6.12 (2.430) | 6.17 (2.420)
Mean Percentage of Daily OFF-time [Mean (Standard Deviation); unit: percentage of daily off time] | 36.86 (13.373) | 38.68 (14.278) | 36.89 (13.490) | 37.47 (13.708)
MDS-UPDRS Part II Total Score [Mean (Standard Deviation); unit: Score on a scale] — Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. Each items had 0-4 ratings, where 0 (normal) to 4 (severe) and score for each was summed to calculate the total scores. The scale range for Part II Total Score was 0-52, with higher scores reflecting greater severity.
  Score on a scale | 13.0 (7.29) | 13.7 (6.65) | 14.1 (7.23) | 13.6 (7.06)
MDS-UPDRS Part III Total Score [Mean (Standard Deviation); unit: Score on a scale] — MDS-UPDRS retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. Each items had 0-4 ratings, where 0 (normal) to 4 (severe) and score for each was summed to calculate the total scores. The scale range for Part III Total Score was 0-136, with higher scores reflecting greater severity.
  Score on a scale | 26.8 (13.99) | 28.7 (13.28) | 27.5 (13.09) | 27.7 (13.46)
PDQ-39 Summary Index [Mean (Standard Deviation); unit: Score on a scale] | 19.97 (13.177) | 20.94 (12.393) | 22.39 (13.115) | 21.07 (12.909)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daily OFF-time During Treatment Period
Description: Reported change from baseline during treatment period which was calculated as follows: Mean for a total of 21 days, consisting of three separate 7-day periods preceding the visits at Week 6, 14 and 26 of the treatment period - Mean for the 7 days preceding the visit at the end of the run-in period. Off-time refers to times when levodopa is not working well, causing worsening symptoms.
Time Frame: From Baseline to Week 26
Population: Full Analysis Set included all randomized participants who received at least 1 dose of the study drug for the treatment period. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 138 | 126 | 122
hours per day | -0.51 (0.167) | -1.11 (0.174) | -1.35 (0.177)
Statistical Analysis 1: Comparison: Placebo vs TVP-1012 1 mg; Test type: Superiority or Other; p = 0.0006, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-1.320 to -0.364] — Estimated Value was reported for the difference between TVP-1012 1mg and Placebo (TVP-1012 1mg - Placebo)
Statistical Analysis 2: Comparison: Placebo vs TVP-1012 0.5 mg; Test type: Superiority or Other; p = 0.0140, ANCOVA; LS Mean Difference = -0.60, 95% CI 2-sided [-1.070 to -0.122] — Estimated Value was reported for the difference between TVP-1012 0.5mg and Placebo (TVP-1012 0.5mg - Placebo)

2. Secondary Outcome: Change From Baseline to Week 26 (LOCF) in Mean Daily OFF-time
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 138 | 126 | 122
hours per day | -0.50 (0.207) | -0.99 (0.217) | -1.40 (0.220)

3. Secondary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II Total Score
Description: MDS-UPDRS retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. Each items had 0-4 ratings, where 0 (normal) to 4 (severe) and score for each was summed to calculate the total scores. The scale range for Part II Total Score was 0-52, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 141 | 132 | 126
Units on a scale | 0.97 (0.408) | -0.30 (0.421) | -0.30 (0.431)

4. Secondary Outcome: Change From Baseline in MDS-UPDRS Part III Total Score
Description: MDS-UPDRS retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. Each items had 0-4 ratings, where 0 (normal) to 4 (severe) and score for each was summed to calculate the total scores. The scale range for Part III Total Score was 0-136, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 140 | 132 | 126
Units on a scale | -3.50 (0.605) | -5.24 (0.623) | -5.65 (0.637)

5. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire-39 (PDQ-39) Summary Index Score
Description: PDQ-39 is a self-administered questionnaire. PDQ-39 comprises of 39 questions, relating to eight key areas (Mobility, Activities of Daily Living, Emotional Well-being, Stigma, Social Support, Cognitions, Communication, and Bodily Discomfort) of health and daily activities, including both Motor and Non-motor symptoms. It is scored on a scale of zero to 100, with lower scores indicating better health and high scores more severe symptoms.
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 138 | 131 | 123
Units on a scale | 2.84 (0.809) | 0.33 (0.829) | -1.00 (0.857)

6. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire-39 (PDQ-39) Each Domain Score
Description: as for outcome 5
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 138 | 131 | 123
Units on a scale
  Mobility | 3.36 (1.515) | -0.64 (1.552) | -2.80 (1.605)
  Activities of Daily Living | 4.42 (1.348) | -1.28 (1.382) | -3.72 (1.429)
  Emotional Well-being | 3.75 (1.295) | -0.01 (1.329) | -0.36 (1.372)
  Stigma | -1.14 (1.161) | -3.28 (1.190) | -2.90 (1.229)
  Social Support | 2.46 (1.043) | 0.60 (1.072) | 1.38 (1.104)
  Cognitions | 1.60 (1.219) | 3.15 (1.252) | 0.69 (1.291)
  Communication | 3.66 (1.107) | 1.59 (1.136) | 2.26 (1.172)
  Bodily Discomfort | 3.36 (1.367) | 2.36 (1.401) | -0.92 (1.449)

7. Secondary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 141 | 133 | 129
Participants
  TEAEs | 71 | 93 | 95
  SAEs | 4 | 10 | 10

8. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Signs Values
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 141 | 133 | 129
Participants
  Temperature (<35.6 °C) | 20 | 21 | 22
  Temperature(>37.7 °C) | 0 | 0 | 1
  Systolic Blood Pressure (<90 mmHg) | 19 | 11 | 27
  Systolic Blood Pressure (>180 mmHg) | 0 | 1 | 1
  Diastolic Blood Pressure(<50 mmHg) | 13 | 16 | 16
  Diastolic Blood Pressure (>100 mmHg) | 4 | 0 | 1
  Pulse (<45 bpm) | 2 | 1 | 1
  Pulse ( >120 bpm) | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With TEAE Related to Body Weight (Weight Decreased)
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 141 | 133 | 129
Participants | 1 | 1 | 2

10. Secondary Outcome: Number of Participants With TEAE Related to Electrocardiograms (ECG) (Sinus Bradycardia)
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 141 | 133 | 129
Participants | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Tests
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Number analyzed (Participants) | 141 | 133 | 129
Participants
  Blood creatine phosphokinase increased | 1 | 1 | 1
  Blood urine present | 0 | 2 | 1
  Gamma-glutamyltransferase increased | 0 | 2 | 0
  Protein urine present | 1 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 1 | 0
  Blood creatine increased | 0 | 1 | 0
  Glucose urine present | 1 | 0 | 0
  Platelet count decreased | 0 | 0 | 1
  Urine ketone body present | 1 | 0 | 0
  White blood cell count decreased | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TVP-1012 0.5 mg | TVP-1012 1 mg
Serious Adverse Events (participants affected / at risk) | 4/141 | 10/133 | 10/129
Other Adverse Events (participants affected / at risk) | 31/141 | 44/133 | 48/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | TVP-1012 0.5 mg (N=133) | TVP-1012 1 mg (N=129)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Disuse syndrome (General disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infective spondylitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | TVP-1012 0.5 mg (N=133) | TVP-1012 1 mg (N=129)
Nasopharyngitis (Infections and infestations) | 13 | 24 | 19
Fall (Injury, poisoning and procedural complications) | 8 | 13 | 17
Contusion (Injury, poisoning and procedural complications) | 2 | 8 | 7
Dyskinesia (Nervous system disorders) | 10 | 11 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.